CLINICAL TRIAL: NCT03235271
Title: Non-Blinded Data Collection Pilot Study of Acute Stroke Using the Brainpulse™
Brief Title: Pilot Study of Acute Stroke Using the Brainpulse™
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMC-1701
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: Severe Ischemic Stroke: Group A will include subjects that present with focal neurological deficits and clinical features consistent with ischemic stroke. Subjects in this group will have a clinical presentation consistent with ischemic stroke and confirmed by radiological imaging. Subjects in this group need to present with an NIHSS score of greater than or equal to 6. Group A is divided into 2 study sub groups of A1 and A2.
  Group A1 are subjects confirmed with acute ischemic stroke secondary to LVO by imaging.
  Group A2 are subjects that present with symptoms of acute ischemic stroke and confirmed to not have an LVO ischemic stroke.
  Interventions: Device: BrainPulse Device
- Group B: Hemorrhagic Stroke: Subjects in this group will present with symptoms similar to Group A. In addition, they will present with clinical symptoms consistent of increased intracranial pressure such as nausea, vomiting, loss of consciousness and severe headache. In order for a subject to be eligible, the hemorrhage will be limited to primarily intracerebral hemorrhage with a minimum volume of 10mL. Subarachnoid hemorrhage and intraventricular hemorrhage may also be present as incidental findings. Since it is unlikely that these subjects proceed for neuro-intervention, they will not have a follow-up BrainPulse recording and they will be exited after completing study procedures.
  Interventions: Device: BrainPulse Device
- Group C: Transient Ischemic Attack: Subjects in this group will present with focal neurological symptoms consistent with stroke. In order for subjects to be eligible for this group, enrollment will need to be within 6 hours of resolution of symptoms along with a confirmation of TIA by treating team. In addition, initial and follow-up radiological imaging needs to show that there are no signs of ischemic stroke or hemorrhage.
  Interventions: Device: BrainPulse Device
- Group D: Non-Stroke Subjects: Group D will include control subjects that do not have an acute stroke. They will be sub-divided into Group D1 and D2.
  Group D1 subjects will be stroke mimics that present with stroke-like symptoms but do not have a diagnosis of stroke or TIA. In order to qualify for this sub group, subjects will also need to show evidence of no stroke on radiological imaging (CT and/or MRI). Diagnoses in this group may include seizure, systemic infection, brain tumor, metabolic disorder, positional vertigo, hemiplegic migraine, encephalopathy, cranial nerve injury, spinal cord injury, brachial/sacral plexus injury, peripheral nerve injury, etc.
  Group D2 subjects will be non-stroke controls that are either patients that present to the hospital for a reason unrelated to stroke and no stroke symptoms or healthy volunteers that are non-clinical visitors or hospital staff. Subjects must have no stroke-like symptoms or suspicion of stroke by the treatment or study team.
  Interventions: Device: BrainPulse Device

INTERVENTIONS:
Device: BrainPulse Device — The BrainPulse is used on a patient's head to non-invasively detect, amplify and capture the skull motion caused by pulsatile cerebral blood flow from the cardiac cycle.
  The BrainPulse consists of a reusable headset that contains the accelerometers used to measure motion caused by pulsatile cerebral blood flow. The system is powered by a rechargeable battery pack. The headset is placed on the subject's head and outputs data to a data collector that forwards the data to the computer. Each accelerometer has an attached tip that makes contact with the subject's head through hair. The headset also includes a photoplethysmograph (PPG) that simultaneously captures the subject's heart-rate information. There is no energy delivered to the brain or subject by these highly sensitive sensors.

SUMMARY:
The aim of this pilot study is to collect data on stroke patients and non-stroke patients or healthy volunteers using the BrainPulse Stroke Monitor. Subject characteristics, diagnostic procedures and clinical outcomes will be documented as part of the data collected to assess the clinical utility of the BrainPulse device. All eligible patients and healthy volunteers will be enrolled and assigned to a study Group based on confirmation of their diagnosis: Acute Ischemic Stroke, Hemorrhagic Stroke, Transient Ischemic Attack or No Stroke. The data collected from the BrainPulse will be compared across the different study groups in an attempt to distinguish stroke from other non-stroke conditions that present with similar symptoms and LVO from non-LVO types of strokes. Further assessments will also be made to evaluate if the BrainPulse can identify the presence of stroke.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, non-blinded, hospital-based study of patients presenting with acute stroke symptoms within 48 hours of symptom onset (last known normal or actual time) as evidenced by radiological imaging. The study will be executed in two parts: Study Phase I and Study Phase II. Each study phase will consist of the same sequence of events and study procedures. The first part of the study is designed to enroll a smaller sample size to evaluate the feasibility of incorporating the BrainPulse device in the Stroke patient care workflow.

Patients will be consecutively recruited and once patients have met eligibility, they will be assigned to one of the four study Groups based on their confirmed clinical diagnosis. Each subject will complete one BrainPulse recording before neuro-intervention and within four hours of IV pharmacologic intervention. All subjects will also complete comprehensive neurological, cognitive and NIH Stroke Scale (NIHSS) assessments. Additionally, Ischemic Stroke subjects (Group A) that receive neuro-intervention will complete one additional, and optional BrainPulse recording along with a neurological exam after intervention. If these procedures have been completed as part of standard of care, the data can be captured directly from the medical records. If such procedures were not conducted as part of hospital's standard of care, they will need to be completed for the purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older
2. Patient undergoes or will undergo radiological imaging (CT/MR) as part of stroke evaluation (n/a for Group D2)
3. Demonstrated at least 1 of the following symptoms (n/a for Group D2):

   1. Hemiparesis, monoparesis, or quadriparesis
   2. Hemisensory deficits
   3. Monocular/binocular visual loss
   4. Visual field deficits
   5. Diplopia
   6. Dysarthria
   7. Facial droop
   8. Ataxia
   9. Vertigo
   10. Aphasia
   11. Severe and sudden onset of headache
   12. Nausea, and/or vomiting
   13. Dizziness
   14. Altered or loss of consciousness
   15. Imbalance/ Incoordination
4. Last known normal or actual time point, whichever is known, since commencement of symptoms < 48 hours prior to enrollment (n/a for Group D2)
5. Consent procedures followed per applicable IRB approvals at site

Exclusion Criteria:

1. Not a candidate for radiological imaging (CT/MR) or angiography (CTA/MRA/DSA) (n/a for Group D2)
2. Patient meets the hospital criteria for brain death
3. Wound or laceration on the head in the area of one of the BrainPulse sensors that would impede use of the BrainPulse device
4. Any serious medical, social or psychological condition that in the opinion of the investigator would disqualify a patient from participation
5. Symptoms due to head trauma
6. IV tPA commenced or completed > 4 hours ago
7. Any neuro-intervention commenced or completed between admission and time of enrollment
8. If does not satisfy the eligibility criteria for groups A, B, C, and D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is expected to enroll up to 289 subjects in total for both parts of the study. During Part I of the study, 40 subjects are expected to be enrolled, of which 20 participants will be assigned to Group A, 5 participants assigned to Group B, 5 participants assigned to Group C, 5 participants assigned to Group D and up to 5 screen failures. In the second part of the study, up to 249 subjects are expected to be enrolled, of which 57 participants will be assigned to Group A1, 57 participants assigned to Group A2, 36 participants assigned to Group D1, and up to 62 participants assigned to group D2, and up to 37 screen failures.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Compare Stroke subject recordings with non-stroke subject recordings | 6 months
  The primary endpoint in Part I of the study is to enroll and record BrainPulse data from 35 eligible subjects who present with classic stroke symptoms and either have a confirmed diagnosis of stroke or no stroke. The BrainPulse device will be used to analyze and compare the differences in signal characteristics between stroke, TIA and control subjects.
Compare differences in signal charactertistics between LVO stroke and all other subjects | 12 months
  BrainPulse signal of all subjects will be analyzed to compare the difference in signal characteristics between LVO stroke and all other subjects enrolled in the study.

SECONDARY OUTCOMES:
Compare Ischemic stroke subject recordings with hemorrhagic stroke or stroke mimic subject recordings | 12 months
  BrainPulse signal will be analyzed to compare the similarity and difference of the BrainPulse signal between hemorrhagic stroke, ischemic stroke subjects or stroke mimics.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Walsh, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - Northwest Community Healthcare, Arlington Heights, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - University of Cincinnati, Department of Emergency Medicine, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided